CLINICAL TRIAL: NCT07331012
Title: The Effects of Upper Extremity Flywheel Exercises on Athletic Skills, Muscle Oxygenation and Physical Fatigue in Adolescent Basketball Players
Brief Title: Effects of Upper Extremity Flywheel Exercises on Skills, Muscle Oxygenation, and Fatigue in Adolescent Basketball
Acronym: Flywheel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Hüseyin Melih Göktuğ Akpulat, MSc Physiotherapist, Istinye University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IstinyeU-EC-25-117
Record Dates: First submitted 2025-12-14; First posted 2026-01-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Physical Fatigue
Keywords: Muscle oxygenation; Upper extremity; Physical fatigue; Flywheel training; Adolescent basketball players; Athletic performance

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: a flywheel training group or a traditional resistance training group. Each group will receive its assigned intervention for 8 weeks, and outcomes will be assessed before and after the intervention period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flywheel Training Group (Experimental): Participants in this group will perform upper extremity eccentric-focused resistance training using a flywheel device. The training program will be conducted for 8 weeks, three sessions per week, in addition to regular basketball training.
  Interventions: Other: Flywheel Exercises
- Traditional Resistance Training Group (Active Comparator): Participants in this group will perform upper extremity resistance training using dumbbells. The training program will be conducted for 8 weeks, three sessions per week, with the same training frequency and duration as the flywheel group, in addition to regular basketball training.
  Interventions: Other: Traditional Resistance Training

INTERVENTIONS:
Other: Flywheel Exercises — Participants perform 8 weeks of upper extremity eccentric resistance exercises using the flywheel device, 3 sessions per week, with progressive load increase over time.
  Arms: Flywheel Training Group
Other: Traditional Resistance Training — Participants perform 8 weeks of upper extremity resistance exercises using dumbbells, 3 sessions per week, with individualized progressive load based on 1 repetition maximum (1RM).
  Arms: Traditional Resistance Training Group

SUMMARY:
This study will investigate the effects of flywheel exercises targeting the upper extremities on athletic performance, muscle oxygenation, physical fatigue, and muscle strength in adolescent basketball players. A total of 36 healthy male adolescent basketball players aged 10-18 years will be included in the study and divided into two groups using stratified randomization: a flywheel exercise group (n=18) and a traditional strength training group (n=18).

Athletic skills will be assessed using the Johnson Basketball Skill Tests (passing test, dribbling test, shooting test), the Basketball Shooting Accuracy Test, and the Functional Shooting Performance Index (FAPI). Upper extremity muscle oxygenation will be measured using near-infrared spectroscopy (NIRS) with a Moxy muscle oxygen meter. Physical fatigue level will be determined using the Modified Borg Scale. Upper extremity muscle strength will be assessed using a Kinvent hand dynamometer and the Seated Single Arm Ball Throw Test. The flywheel group will undergo eccentric weight flywheel exercises three times a week for eight weeks. The traditional strength training group will follow a strength training program using dumbbells for the same duration and frequency. All assessments will be conducted before and after the training program.

DETAILED DESCRIPTION:
Adolescence is a critical period in which athletic performance and musculoskeletal adaptations develop rapidly. In sports that actively utilize the upper extremities, such as basketball, strength, coordination, and fatigue tolerance directly affect performance. In recent years, flywheel exercise systems, which allow for eccentric loading, have emerged as an effective training method for improving muscle strength and neuromuscular adaptations. However, scientific evidence regarding the effects of these systems on adolescent athletes is limited. This study was planned to investigate the effects of flywheel exercises targeting the upper extremities on athletic performance, muscle oxygenation, and physical fatigue in adolescent basketball players. The study will be conducted using a randomized controlled design, with participants divided into two groups: a flywheel exercise group and a traditional strength training group. Both groups will receive a structured upper extremity strength training program of equal duration and frequency. Throughout the study, all participants will continue their routine basketball training; only the strength training method applied will differ between the groups. Assessments will be conducted before and after the training program, and intra-group and between-group changes will be analyzed. The findings are expected to provide important information about the applicability of flywheel exercises in adolescent athletes and their potential effects on performance.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer male basketball players aged 10-18 who have played basketball for at least one year,
* Who have regularly attended training sessions for the past 6 months,
* Who do not have an injury that would restrict their participation in training will be included in the study.

Exclusion Criteria:

* Those who have undergone upper extremity surgery within the last year
* Those with neurological, cardiovascular, respiratory, or metabolic diseases (e.g., epilepsy, heart disease, asthma, diabetes, etc.)
* Those who have sustained any upper extremity musculoskeletal injury within the last year

Ages: 10 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Basketball-Specific Skill Performance | Baseline and after 8 weeks of training
  Basketball-specific skills will be assessed using the Johnson Basketball Skill Tests (passing, dribbling, and shooting tests), the Basketball Shooting Accuracy Test, and the Functional Throwing Performance Index (FTPI). Higher scores indicate better basketball-specific skill performance."
Muscle Oxygenation | Baseline and after 8 weeks of training
  Upper extremity muscle oxygenation will be assessed using near-infrared spectroscopy (NIRS) with a Moxy muscle oxygen monitor placed over the biceps brachii muscle during basketball-specific performance tasks. Higher oxygen saturation percentages indicate better muscle oxygenation.
Physical Fatigue | Baseline and after 8 weeks of training
  Perceived physical fatigue will be assessed using the Modified Borg Rating of Perceived Exertion (RPE) Scale, which ranges from 0 (no fatigue) to 10 (maximal fatigue). Higher scores indicate greater perceived physical fatigue.

SECONDARY OUTCOMES:
Upper Extremity Isometric Muscle Strength | Baseline and after 8 weeks of training
  Upper extremity isometric muscle strength will be assessed using a Kinvent handheld dynamometer. Measurements will include shoulder and elbow muscles. Strength will be recorded in kilograms or Newtons. Higher values indicate greater isometric strength.
Upper Extremity Explosive Strength | Baseline and after 8 weeks of training
  Upper extremity explosive strength will be evaluated using the Seated Single-Arm Medicine Ball Throw Test. Participants throw a medicine ball as far as possible from a seated position. Distance of the throw will be recorded in centimeters. Higher values indicate greater explosive strength.

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Melih Goktug Akpulat, Principal Investigator — Istinye University
Locations (1):
- Iğdır Youth and Sports Provincial Directorate - Kazım Karabekir Sports Hall, Iğdır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the small sample size, the involvement of adolescent participants, and data protection and confidentiality considerations. Data will be used only for the purposes defined in the study protocol.

REFERENCES:
- [Background] Younes-Egana O, Mielgo-Ayuso J, M Stojanovic MD, Bird SP, Calleja-Gonzalez J. Effectiveness of Eccentric Overload Training in Basketball Players: A Systematic Review. J Hum Kinet. 2023 Jul 15;87:243-257. doi: 10.5114/jhk/167469. eCollection 2023 Jul. PMID 37559764